CLINICAL TRIAL: NCT06033638
Title: Agreement and Inter-rater Reliability of Video Documented PBS-Score - An International Cross-sectional Multicenter Study
Brief Title: Video Documented PBS-Score in Children With Clubfoot
Acronym: PEVA
Status: Completed | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Eva Weidenhielm-Brostrom, Manager, Region Stockholm
Other Study IDs: K 2022-10475
Record Dates: First submitted 2023-05-10; First posted 2023-09-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Clubfoot; PBS
MeSH Terms: conditions — Clubfoot | interventions — Organ Dysfunction Scores

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Score assessment — PBS Score
  Other Names: PBS-score, video evaluation, PROM

SUMMARY:
Evaluate agreement and inter-rater reliability of PBS-score assessments based on video documented material.

DETAILED DESCRIPTION:
120 children with idiopathic clubfoot will be included from four different countries 30 patients from each participating center. Inclusion criteria include: age 4-14 years, diagnosis of idiopathic clubfoot, ability to walk 10 m repeatedly, and ability to communicate verbally (and in writing for caregivers) in Swedish, English, Portuguese, Urdu, or Pashto. All items of the PBS-score will be documented using video recordings. Six to eight senior orthopedic surgeons will score a total of 90 children each, not the children from their center of employment, according to the PBS-score based on videos. Collaborating centers include Karolinska University Hospital, Sweden, Hospital Pequeno Príncipe, Brazil, and Hayatabad Medical Complex, Orthopaedic Unit, Peshawar, Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* Clubfoot

Exclusion Criteria:

-

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children born with clubfoot
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
PBS Score agreement and inter-rater reliability | 1 year
  PBS Score is a tool to grade the severity of clubfoot recurrence in the walking child, and was proposed to serve as an instrument to guide treatment. The sum of all points for all signs is scored between 7 and 18.

CONTACTS AND LOCATIONS:
Overall Officials: Eva W Broström, Professor, Principal Investigator — Astrid Lindgren Children´s Hospital
Locations (1):
- Astrid Lindgren Children´s Hospital, Stockholm, Region Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No